CLINICAL TRIAL: NCT06616831
Title: Development of At-Home Transcutaneous Auricular Vagus Nerve Stimulation for Post-Stroke Rehabilitation
Brief Title: At-Home taVNS - Stroke Rehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00137256
Record Dates: First submitted 2024-08-12; First posted 2024-09-27 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Remote Transcutaneous Auricular Vagal Nerve Stimulation Paired with Task Specific Training (Experimental): Task-specific training (TST) paired with EMG activated Transcutaneous Auricular Vagal Nerve Stimulation (taVNS) three times a week for two weeks in an At-Home setting.
  Interventions: Device: Remote Transcutaneous Auricular Vagal Nerve Stimulation Paired with Task-Specific Training

INTERVENTIONS:
Device: Remote Transcutaneous Auricular Vagal Nerve Stimulation Paired with Task-Specific Training — Each participant will complete 2 weeks, 3 times per week, task-specific training paired with transcutaneous auricular vagal nerve stimulation.

SUMMARY:
Early evidence suggests the benefits of post-stroke motor rehabilitation may be enhanced by applying electrical stimulation to the ear. This study aims to test the new approach of pairing ear stimulation with motor rehabilitation in the home setting in stroke survivors with upper limb motor function deficits.

DETAILED DESCRIPTION:
This study seeks to advance prior research conducted here at MUSC exploring the use of transcutaneous auricular vagus nerve stimulation (taVNS) paired with motor rehabilitation to improve motor function post-stroke. Early evidence from a recently completed NIH-funded, clinical trial suggests that our new approach of delivering electrical stimulation to the ear at the same time as motor rehabilitation double the clinical benefits of motor rehabilitation. These benefits are due in part to a facilitation of neuroplasticity caused by activating the auricular branch of the vagus nerve.

This project takes this approach one step further, moving it into the home in combination with telerehabilitation in order to make this technology more accessible to individuals in rural and remote areas. In order to accomplish this, investigators will a) conduct lab-based testing and validation of the stimulation triggering sensors for at-home use, and b) determine the safety, feasibility, and acceptability of at-home taVNS in five stroke survivors with unilateral upper limb motor deficits.

Investigators hypothesize that our lab-based validation will facilitate an optimized home intervention. Furthermore, investigators hypothesize taVNS will be safe and feasible to self-administer in the at-home setting. Lastly, investigation will help elucidate any challenges that may occur as investigators begin to expand this technology into future larger trials

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old with an ischemic or hemorrhagic stroke that occurred ≥6 months prior;
* Ability to give consent;
* Unilateral limb (left or right) weakness with Fugl Meyer-Upper Extremity Scale score of 19-53/60 points which indicates adequate arm/hand use for rehabilitation tasks;
* active wrist flexion/extension ≥10° with active abduction/extension of thumb and at least 1 digit ≥10° to further assure ability to participate in rehabilitation tasks;
* Passive range of motion in affected shoulder, elbow and wrist within 20 degrees of normal values.

Exclusion Criteria:

* Other concomitant neurological disorders affecting upper extremity motor function;
* Presence of Dysphagia or aspiration difficulties;
* Prior injury to vagus nerve;
* Pregnancy;
* Documented history of dementia before or after stroke;
* Documented history of uncontrolled depression or psychiatric disorder either before or after stroke which could affect their ability to participate in the experiment;
* Uncontrolled hypertension;
* Botox injections within 4 weeks of the first day of rehabilitation therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility through dropout rates | 2 weeks
  Dropout rates will be assessed over the course of the study.
Safety of stimulation | 2 weeks
  Any side effects or adverse events will be assessed.
Compliance | 2 weeks
  Compliance with study procedures will be assessed every study visit.
Subjective ratings of feasibility. | 2 weeks
  Feasibility will be assessed with subjective ratings on subject's ability to complete study procedures at home.

SECONDARY OUTCOMES:
Compliance with at-home sessions | 2 weeks
  The total number of completed at-home sessions will be measured. The total stimulation duration completed within each session. Benchmarks of >80% total motor rehabilitation sessions completed, and 45 minute in-session duration will be the feasibility cutoffs for the analysis.
Motor Function | 2 weeks
  Motor function will be assessed in-person at baseline and at the end of the two-week intervention using the Fugl-Meyer Assessment (FMA).

CONTACTS AND LOCATIONS:
Overall Officials: Bashar Badran, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badran BW, Peng X, Baker-Vogel B, Hutchison S, Finetto P, Rishe K, Fortune A, Kitchens E, O'Leary GH, Short A, Finetto C, Woodbury ML, Kautz S. Motor Activated Auricular Vagus Nerve Stimulation as a Potential Neuromodulation Approach for Post-Stroke Motor Rehabilitation: A Pilot Study. Neurorehabil Neural Repair. 2023 Jun;37(6):374-383. doi: 10.1177/15459683231173357. Epub 2023 May 20. PMID 37209010